CLINICAL TRIAL: NCT07079566
Title: Effect of Primal Reflex Release Technique on Pain and Function in Plantar Fasciitis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC_02002
Record Dates: First submitted 2025-07-02; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Planter Fasciitis

STUDY DESIGN:
Intervention Model Description: In this parallel assignment randomized controlled trial, participants diagnosed with plantar fasciitis were randomly allocated into two groups: the experimental group and the control group. The experimental group received Primal Reflex Release Technique (PRRT) along with routine physiotherapy care, while the control group received only routine standard care including stretching and strengthening exercises. The intervention duration was 3 weeks, with baseline assessments conducted in the first week and post-intervention assessments at the end of the third week. Randomization was achieved through non-probability purposive sampling followed by simple random allocation. The primary aim was to assess changes in pain intensity and foot function using the Numeric Pain Rating Scale (NPRS) and Foot Function Index (FFI), respectively. Data analysis included pre- and post-intervention comparisons to determine the effectiveness of PRRT.
Who Masked: Participant
Masking Description: In this randomized controlled trial, a single-masked (assessor-blinded) design was used. Participants were randomly assigned to either the experimental group receiving the Primal Reflex Release Technique (PRRT) or the control group receiving conventional treatment. Due to the hands-on and physical nature of the PRRT intervention, it was not feasible to blind participants or treating therapists. However, to reduce the risk of detection and measurement bias, the outcome assessors responsible for evaluating the pre- and post-intervention scores were blinded to the group allocation. These assessors collected data using validated outcome measures, including the Numeric Pain Rating Scale (NPRS) and Foot Function Index (FFI). They were not involved in the treatment sessions and were unaware of which participants received which intervention. so it means thatthis blinding procedure was designed to maintain objectivity in data collection and enhance the internal validity of the study results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primal Reflex Release Technique (PRRT) Group A (Experimental): Participants in this group will receive the Primal Reflex Release Technique (PRRT), a hands-on manual therapy based on the principle of modulating overactive primal reflexes believed to contribute to chronic musculoskeletal pain and dysfunction. The intervention is designed to target reflexive neuromuscular responses to reduce muscle guarding and pain. The PRRT sessions will be administered by a trained physiotherapist over a 3-week period, with three sessions per week, totaling nine sessions. Each session will last approximately 20-30 minutes. The technique includes procedures like sternocleidomastoid release, startle reflex inhibition, and skin stretch methods. The aim is to reduce plantar fascia tension by addressing upstream reflexive tension patterns. All participants will be assessed pre- and post-intervention using the Numeric Pain Rating Scale and Foot Function Index to evaluate changes in pain and functional ability.
  Interventions: Behavioral: Primal Reflex Release Technique (PRRT)he Primal Reflex Release Technique (PRRT) is a hands-on, non-invasive therapeutic approach designed to deactivate overactive protective reflexes believed to contr
- Conventional Physiotherapy Group B (Active Comparator): Participants in this group will receive conventional physiotherapy treatment commonly used for plantar fasciitis management. This includes static stretching of the plantar fascia and Achilles tendon, strengthening exercises for intrinsic foot muscles, heel cord stretches, ice therapy, footwear advice, and patient education. The treatment will also be provided over 3 weeks, with sessions scheduled three times per week for a total of nine sessions, each lasting 20-30 minutes. This standard care group serves as the control arm to evaluate the comparative effectiveness of the Primal Reflex Release Technique. All participants in this group will undergo pre- and post-intervention assessment using the Numeric Pain Rating Scale (NPRS) and the Foot Function Index (FFI) to measure changes in pain levels and foot-related functional limitations.
  Interventions: Behavioral: Conventional Physiotherapy Treatment This reflects the standard care or routine treatment used as a comparison in your randomized controlled trial on plantar fasciitis. Let me know if your control gr

INTERVENTIONS:
Behavioral: Primal Reflex Release Technique (PRRT)he Primal Reflex Release Technique (PRRT) is a hands-on, non-invasive therapeutic approach designed to deactivate overactive protective reflexes believed to contr — The Primal Reflex Release Technique (PRRT) is a non-invasive, manual therapy that targets specific neurogenic reflex points to reduce muscle tension, pain, and dysfunction. It works by modulating the autonomic nervous system to interrupt hyperactive primal reflexes such as withdrawal and startle reflexes, which are often involved in chronic musculoskeletal pain conditions like plantar fasciitis. In this study, PRRT was applied to participants in the experimental group over a 3-week period, consisting of multiple sessions per week. Each session included a series of gentle manual techniques such as the sternocleidomastoid (SCM) release, startle reflex inhibition, and positional reflex modulation. These techniques aim to reset the body's reflex-driven pain responses and promote functional mobility. PRRT was performed by trained physiotherapists following a standardized protocol to ensure consistency throughout the study.
  Arms: Primal Reflex Release Technique (PRRT) Group A
Behavioral: Conventional Physiotherapy Treatment This reflects the standard care or routine treatment used as a comparison in your randomized controlled trial on plantar fasciitis. Let me know if your control gr — The control group in this randomized controlled trial received standard conventional physiotherapy treatment for plantar fasciitis. This treatment protocol consisted of traditional evidence-based physiotherapy interventions commonly used in clinical practice. Participants received supervised sessions including static and dynamic stretching exercises targeting the plantar fascia, Achilles tendon, and calf muscles. In addition, the intervention included modalities such as cryotherapy (application of ice packs), ultrasound therapy for soft tissue healing, and patient education on activity modification, proper footwear, and home exercise programs.
  The conventional treatment was administered for 3 sessions per week over a period of 3 weeks. Each session lasted approximately 30 to 40 minutes. The objective of this intervention was to reduce inflammation, relieve pain, and improve foot function through mechanical and thermal means, without involving neuromuscular reflex reprogramming. This a
  Arms: Conventional Physiotherapy Group B

SUMMARY:
The plantar fascia at the foot bottom causes pain and inflammation which affects this thick tissue that runs from heel bone to toe. This condition stands as the main source of heel pain and produces intense stabbing sensations which become noticeable in the morning and during periods of rest. The foot pain generally reduces when a foot becomes active but it often resurfaces after standing or being active for prolonged periods of time(1).

Plantar fasciitis occurs as a frequent problem which affects 10% of people worldwide during their lifespans. Annual plantar fasciitis cases in adults reach 1% within the United States while medical care is provided to over 2 million people annually. Research shows that plantar fasciitis affects a similar proportion of people in the United Kingdom during their lifetime at about 10%(2). The prevalence rate for plantar fasciitis in Pakistan remains unclear because studies show that 4.72% of housewives in Lahore experience the condition. Plantar fasciitis represents a widespread foot condition worldwide since it affects numerous population groups based on these statistical reports(3).

The main symptom of plantar fasciitis manifests as heel pain that feels either sharp and burning and stabbing. Heel pain reaches its highest intensity during the morning after a person wakes up because of the initial foot movements. Heel pain intensifies when maintaining a resting position but subsides as the affected person becomes active. The medical condition becomes worse due to high amounts of physical activity that results in daily foot pain(4).

Many patients report foot sensitivity combined with swellings that develop either in the heel zone or beneath the foot arch. The heel area tends to experience pain PRT establishes an efficient pain management strategy through its ability to treat nervous system dysfunctions which generate chronic pain and inflammatory conditions. PRRT improves health outcomes along with reducing treatment duration while it substantially enhances the life quality of people who experience prolonged pain. The body's natural pain relievers activate through non-invasive movements in Primal Reflex Release Technique which makes this method important for treating plantar fascitis.Through reflex activation PRT activates natural pain-relieving mechanisms of the brain thus leading to substantial pain reduction and improved inflammation levels. The direct intervention on pain-causing nerve dysfunctions resulting from chronic pain through PRT activates healthy nervous system operations(25).

The best results from PRT emerge when patients use it together with physical therapy along with stretching and strengthening therapeutic exercises. The therapy presents both gentle nature and noninvasive methods with combined benefits of using little to no medical drugs or special devices. The therapy serves alongside multiple therapeutic approaches for treating enduring pain issues and inflammatory conditions of the back, neck, and head along with fibromyalgia and arthritis and tendinitis and plantar fasciitis. The therapy provides therapeutic benefits in neurological medical fields which assist patients with sciatica and neuropathy complications and Parkinson's disease conditions.

DETAILED DESCRIPTION:
The Primal Reflex Release Technique (PRRT) was used to treat Medial Tibial Stress Syndrome (MTSS) in NCAA Division I cheerleaders. Three male and two female participants, with a mean age of 20 ± 1.4 years, who had been diagnosed with Type II MTSS, received PRRT treatment. The research indicated both immediate pain relief after a single treatment session and functional enhancement after an average of 4.2 (± 0.84) sessions over 15.4 (± 5.86) days, all without any imposed training pauses. Patient outcomes from PRRT showed lasting improvements during both the initial follow-up and the two-week check-up, indicating the effectiveness of this method for MTSS patients. The study suggests that PRRT shows promise as a non-invasive therapy for the effective management of stress-related tibial pain in athletic populations (29).

Current literature on plantar fasciitis syndrome (PFS) treatment using manual physiotherapy is limited. Therefore, a randomized controlled trial was conducted by Khammas et al. (2024) to evaluate the efficacy of manual physiotherapy in altering plantar fascia morphology, including changes in the thicknesses of the central fascial portion (CFP) and the key fascial portion (KFP), pain levels, and foot function in PFS patients. The participants were divided into three groups: Group A (40 PFS patients receiving manual physiotherapy), Group B (42 PFS patients receiving no intervention), and Group C (40 healthy controls matched for age, gender, and BMI). Results showed a significant increase in plantar fascia thickness in Groups A and B (P < 0.001). However, Group A showed significant improvements in plantar fascia thickness, echogenicity, CFP thickness (P < 0.001), pain reduction, and functional performance-particularly in acute cases of PFS (30).

The foot and ankle play essential roles in locomotion, functioning as shock absorbers, allowing adaptation to uneven surfaces, and providing stability. Dysfunction in this region can contribute to issues involving the knee, hip, spine, and can lead to recurrent stress fractures, plantar fasciitis, and tibial stress syndromes. These dysfunctions need to be addressed through biomechanical and neuromuscular reflexive approaches. The Primal Reflex Release Technique (PRRT) is of interest due to its influence on involuntary reflexive responses. PRRT helps reset dysfunctional neuromuscular patterns to alleviate pain and improve function in conditions such as plantar fasciitis and MTSS, making it a promising, non-invasive intervention for both athletes and chronic sufferers of foot and lower limb pain (31).

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years and of both genders.
* Diagnosed with Plantar Fasciitis by a healthcare professional
* Experiencing heel pain or pain at the bottom of the foot for at least 3 months or more than 3 months
* Patient with acute or chronic planter fasciitis Positive windless test.
* Pain with walking or dorsiflexion of the toes, especially in the morning Willing to adhere to the study protocol

Exclusion Criteria:

* Participants were excluded if they have any of the following: Previous surgery for Plantar Fasciitis
* Systemic inflammatory conditions (e.g., rheumatoid arthritis) Pregnancy
* Neurological disorders affecting the lower limbs Other foot pathologies (e.g., tarsal tunnel syndrome)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity using Numeric Pain Rating Scale | Baseline and after 3 weeks of intervention
  The Numeric Pain Rating Scale (NPRS) is an 11-point scale used to assess the intensity of pain. Patients rate their current pain from 0 (no pain) to 10 (worst imaginable pain). This study assesses change in NPRS scores from baseline to post-intervention. The tool is highly reliable (r = 0.95-0.98) and valid (r = 0.85-0.95) for clinical use.

SECONDARY OUTCOMES:
Change in Foot Function using Foot Function Index (FFI) | Baseline and after 3 weeks of intervention ❗️Summary of Fixes: All repeated NPRS entries were consolidated into one primary measure. The "Time Frame: 3" issue was corrected by clearly stating "Baseline and after 3 weeks of intervention". The secondary
  The Foot Function Index (FFI) is a self-reported questionnaire designed to measure foot pain, disability, and activity limitation. It includes 23 items across 3 subscales (pain, disability, and activity limitation), each scored from 0 to 10. The total score is expressed as a percentage, with higher scores indicating greater disability. This outcome assesses the change in FFI scores before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shamaila yaqub, MS OMPT, Principal Investigator — riphah international university gulberg green campus islamabad
Locations (1):
- Lady reading hospital MTI peshawar, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No